CLINICAL TRIAL: NCT01293435
Title: Observational Study to Assess Clinical Management Patterns in Patients With Hospitalised Community-Acquired Pneumonia (CAP) or Complicated Skin and Skin Structure Infections (cSSSI)
Brief Title: Study Evaluating Management of Patients With Community-Acquired Pneumonia (CAP) or Complicated Skin Infections
Acronym: REACH
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-IEU-DUM-2010/1
Record Dates: First submitted 2011-02-06; First posted 2011-02-10 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Community Acquired Pneumonia (CAP); Complicated Skin and Skin Structures Infections (cSSSI)
Keywords: Community Acquired Pneumonia (CAP); Complicated Skin and Skin Structures Infections (cSSSI); Complicated Skin and Soft Tissues Infections (cSSTI); Antibiotics; Infection management; Use of Resources; MRSA; PRSP
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study will collect real-life data from patients with community acquired pneumonia (CAP) OR complicated skin and skin structure infections (cSSSI) to assess the burden of the disease, review the treatment pathways, evaluate how health resources are used and identify any areas of unmet medical needs. The aim of the study is to compare how patients who are admitted to hospital with CAP or cSSSI are managed across Europe. This will be done by collecting data to understand the patient and disease characteristics, current practice of treatment, and outcomes for the patient. Overall 4000 patients will be recruited from 10 European countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised with CAP or cSSSI

  1. CAP: Radiographically-confirmed bacterial pneumonia AND Requiring treatment with IV antimicrobials as start-up therapy
  2. cSSSI: Affecting deeper soft tissue and/or requiring significant surgical intervention or developing an abcess/ulcer/cellulitis in a lower limb AND Having at least two local signs and one systemic sign of cSSS AND Treatment with antimicrobials

Exclusion Criteria:

* Patients already participating in clinical trials or any other interventional study.

  1. CAP: CAP suitable for outpatient therapy with an oral antimicrobial agent.
  2. cSSSI: Uncomplicated SSSI. Skin and skin-structure infections with a high cure rate after surgical incision alone or after aggressive local skin care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18, diagnosed with community acquired pneumonia or complicated skin and skin structure infection hospitalised between 2010-12-01 and 2011-01-31.
Sampling Method: Probability Sample
Enrollment: 4035 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with infection resolution reaching clinical stability, as a measure of effectiveness | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).
Number of patients reaching clinical stability, as a measure of effectiveness | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).
Number of patients death, as a measure of clinical failure | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).
Number of patients with infection recurrence, as a measure of clinical failure | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).
Number of patients requiring change in antibiotic, as a measure of clinical failure | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).

SECONDARY OUTCOMES:
Number of patients hospitalized with CAP or cSSSI, in each type of hospital and department, as a descriptive measure of burden of disease, and patient flow. | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31.
Number and type of diagnostic tests, as measure of use of resources | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).
Type of medications used, as measure of use of resources | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).
Duration of hospitalisation, as measure of use of resources | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).
Number of patients requiring ICU / isolation / mechanical ventilation / complications, as measure of use of resources | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).
No. patients infected with MR-Staphylococcus aureus in cSSSI, or with PR-Streptococcus pneumoniae in CAP, not responding to antibiotic treatment, as measure of prevalence of resistant strains and of incidence of associated clinical failure | Retrospective. Outcome measures will be determined in patients hospitalized between 2010-12-01 and 2011-01-31, from the date of hospitalization, up to the date of hospital discharge (2011-02-28 at the latest).

CONTACTS AND LOCATIONS:
Locations (163):
- Belgium (11):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Dinant
  - Research Site, Edegem
  - Research Site, Godinne
  - Research Site, Hasselt
  - Research Site, Liège
  - Research Site, Mons
  - Research Site, Montigny-le-Tilleul
- France (51):
  - Research Site, Alençon
  - Research Site, Amboise
  - Research Site, Amiens
  - Research Site, Bayonne
  - Research Site, Bergerac
  - Research Site, Briançon
  - Research Site, Brive-la-Gaillarde
  - Research Site, Cahors
  - Research Site, Cayenne
  - Research Site, Chambéry
  - Research Site, Chauny
  - Research Site, Cognac
  - Research Site, Colombes
  - Research Site, Compiègne
  - Research Site, Creil
  - Research Site, Decazeville
  - Research Site, Denain
  - Research Site, Dunkirk
  - Research Site, Eaubonne
  - Research Site, Évreux
  - Research Site, Fécamp
  - Research Site, Hyères
  - Research Site, La Tronche
  - Research Site, Lagny-sur-Marne
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Le Mans
  - Research Site, Lens
  - Research Site, Libourne
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Metz
  - Research Site, Montdidier
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pontarlier
  - Research Site, Rethel
  - Research Site, Saint-Aubin-lès-Elbeuf
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Dié
  - Research Site, Saint-Hilaire-du-Harcouët
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saint-Quentin
  - Research Site, Saintes
  - Research Site, Salon-de-Provence
  - Research Site, Strasbourg
  - Research Site, Tarbes
  - Research Site, Toul
  - Research Site, Tulle
  - Research Site, Vendôme
  - Research Site, Vesoul
- Germany (8):
  - Research Site, Ulm, Baden-Wurttemberg
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Dortmund, North Rhine-Westphalia
  - Research Site, Paderborn, North Rhine-Westphalia
  - Research Site, Kiel, Schleswig-Holstein
  - Research Site, Lübeck, Schleswig-Holstein
  - Research Site, Berlin, State of Berlin
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Crete
  - Research Site, Larissa
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Italy (30):
  - Research Site, S.G. Rotondo, Foggia
  - Research Site, Rozzano, Milano
  - Research Site, Pietra Ligure, Savona
  - Research Site, Borgo Roma, Verona
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Chieti
  - Research Site, Cuneo
  - Research Site, Enna
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Latina
  - Research Site, Lodi
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Pesaro
  - Research Site, Pisa
  - Research Site, Reggio Calabria
  - Research Site, Roma
  - Research Site, Sassari
  - Research Site, Savona
  - Research Site, Siena
  - Research Site, Torino
  - Research Site, Varese
- Netherlands (9):
  - Research Site, Harderwijk, Gelderland
  - Research Site, Breda, North Brabant
  - Research Site, Nieuwegein, Utrecht
  - Research Site, Breda
  - Research Site, Groningen
  - Research Site, Leiden
  - Research Site, Nijmegen
  - Research Site, Utrecht
  - Research Site, Zoetermeer
- Portugal (7):
  - Research Site, Amadora
  - Research Site, Lisbon
  - Research Site, Penafiel
  - Research Site, Portimão
  - Research Site, Torres Novas
  - Research Site, Viana do Castelo
  - Research Site, Vila Nova de Gaia
- Spain (14):
  - Research Site, Terrassa, Barcelona
  - Research Site, Santiago de Compostela, Coruna
  - Research Site, Vigo, Pontevedra
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
- Turkey (Türkiye) (18):
  - Research Site, Bolu, Abant
  - Research Site, Izmir, Balova
  - Research Site, Ankara, Be?evler
  - Research Site, Ankara, Besevler
  - Research Site, Ankara, Bilkent
  - Research Site, Izmir, Bornova
  - Research Site, ?zmir, Bozyaka
  - Research Site, Istanbul, Capa
  - Research Site, Istanbul, Cerrahpasa
  - Research Site, Ankara, Dskapi
  - Research Site, Antalya, Dumlupinar Mevkii
  - Research Site, ?stanbul, Kartal
  - Research Site, Istanbul, Mraniye
  - Research Site, Bursa, Nilfer
  - Research Site, Samsun, Ondokuz Mayıs
  - Research Site, Eskiehir, Osmangazi
  - Research Site, Ankara, S?hhiye
  - Research Site, Ankara, Sihhiye
- United Kingdom (9):
  - Research Site, Aintree
  - Research Site, Blackpool
  - Research Site, Edinburgh
  - Research Site, Hull
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, Middlesbrough
  - Research Site, Newcastle
  - Research Site, Winchester

REFERENCES:
- [Derived] Garau J, Blasi F, Medina J, McBride K, Ostermann H; REACH study group. Early response to antibiotic treatment in European patients hospitalized with complicated skin and soft tissue infections: analysis of the REACH study. BMC Infect Dis. 2015 Feb 19;15:78. doi: 10.1186/s12879-015-0822-2. PMID 25879713
- [Derived] Blasi F, Ostermann H, Racketa J, Medina J, McBride K, Garau J; REACH study group. Early versus later response to treatment in patients with community-acquired pneumonia: analysis of the REACH study. Respir Res. 2014 Jan 22;15(1):6. doi: 10.1186/1465-9921-15-6. PMID 24450444
- [Derived] Blasi F, Garau J, Medina J, Avila M, McBride K, Ostermann H; REACH study group. Current management of patients hospitalized with community-acquired pneumonia across Europe: outcomes from REACH. Respir Res. 2013 Apr 15;14(1):44. doi: 10.1186/1465-9921-14-44. PMID 23586347